CLINICAL TRIAL: NCT01433835
Title: Safety and Pharmacokinetics of Single Oral Doses of MBX-400 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Microbiotix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-001
Record Dates: First submitted 2011-09-11; First posted 2011-09-14 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Adult Subjects
Keywords: Cytomegalovirus; Antiviral; Safety; Healthy
MeSH Terms: interventions — cyclopropavir; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- MBX-400 (Experimental)
  Interventions: Drug: MBX-400

INTERVENTIONS:
Drug: MBX-400 — Capsule(s) for oral administration as a single dose. Planned doses include: 35, 100, 350, 700, 1000 and 1350 mg.
  Other Names: ZSM-I-62; NSC D745998; Cyclopropavir (CPV); (Z)-9-{[2,2-bis-(hydroxymethyl)cyclopropylidene] methyl}guanine
  Arms: MBX-400
Other: Placebo — Capsule(s) for oral administration as a single dose. Planned doses include: 35, 100, 350, 700, 1000 and 1350 mg.
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and pharmacokinetics following a single oral dose of MBX-400.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV; herpesvirus 5), a member of the betaherpesvirus subgroup, occurs as a benign infection in the majority of humans, with a 90% prevalence in the adult population1. However, CMV infection continues to be a major cause of morbidity and mortality in immunosuppressed patients, particularly recipients of solid organ or bone marrow transplants. CMV is also known for its association with severe blinding retinitis, pneumonia and gastrointestinal inflammation in AIDS patients. However, with the successful introduction of HAART (highly active anti-retroviral therapy), the problem of CMV infection in AIDS patients has decreased substantially. CMV remains the most important cause of congenital viral infection in the United States, and CMV infection of neonates is associated with deafness, mental retardation and mortality. In addition, CMV is a suspected pathogenic agent in cardiovascular disease and can persist in large-vessel endothelial cells and infect all cell types involved in cardiovascular lesions. CMV has been implicated in the restenosis of diseased coronary arteries following angioplasty and has been associated with myocarditis. In severely immunocompromised patients with CMV infection, prolonged antiviral therapy is often necessary, which increases the risk of resistant viruses. Currently available therapy has limitations that preclude their long-term use including toxicity, poor oral bioavailability and the development of drug-resistant strains. MBX-400 is a nucleoside analog that is structurally related to ganciclovir and acyclovir and is being developed for the possible use in the prevention and/or treatment of CMV. MBX-400, has been shown to be a potent inhibitor of viral DNA synthesis and therefore may be useful in treating and/or preventing CMV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 65 years of age
2. Females must be surgically-sterilized or post-menopausal (defined as at least 1 year since last menses with follicle stimulating hormone (FSH) level indicating subject is post-menopausal)
3. Males must have undergone vasectomy
4. Able to understand study requirements, agrees to participate in the study and willing and able to provide informed consent (using an informed consent form in a language in which the subject is fluent)
5. Willing and able to stay in a clinical facility for up to 7 days
6. BMI of 18 to 32 kg/m2
7. Non-smoker or former smoker or user of nicotine-containing products (defined as someone who smoked or used nicotine-products one or more times a week for at least one month) who has not smoked for at least 3 months and has not used nicotine-containing products for at least 1 month and is willing to abstain from nicotine-containing products during the study
8. Has adequate venous access
9. Willing to abstain from alcohol and illicit drugs during the study

Exclusion Criteria:

1. Participation in another clinical trial within 3 months of screening
2. Unwilling to comply with study procedures or cooperate with study personnel.
3. Donated blood or had significant blood loss (greater than 1 unit) within 3 months of screening
4. History of any of the following

   * Human immunodeficiency virus (HIV), cytomegalovirus (CMV), hepatitis B or hepatitis C infection
   * Alcohol or drug abuse
   * Anemia or bleeding disorders
   * Gastrointestinal disorders
   * Chronic illness
   * Regular medication use (prescription, over-the-counter or herbal; defined as more than once per week; except multivitamins) or use of medication (except multivitamins) within 1 week of screening.
   * Recent illness requiring treatment within 1 month of screening
   * History of renal failure or renal insufficiency
5. Clinically significant abnormal electrocardiogram (e.g., abnormal rhythm, abnormal intervals)
6. Clinically significant results of hematology, chemistry, coagulation studies or urinalysis, including, but not limited to the following:

   * White blood cell count, red blood cell count or platelet count less than the lower limit of normal or greater than 1.5 times the upper limit of normal
   * Hemoglobin or hematocrit less than the lower limit of normal or greater than the upper limit of normal
   * Alanine aminotransferase and aspartate aminotransferase greater than the upper limit of normal
   * Prothrombin, partial thromboplastin time or international normalized ratio greater than 1.5 times the upper limit of normal
   * Abnormal electrolyte values (i.e., sodium, potassium, carbon dioxide/bicarbonate, chloride and/or calcium outside of the reference range)
   * Urinalysis showing presence of red blood cells, protein or microalbumin
   * Cotinine level indicative of nicotine use
   * Positive test for any drug of abuse on urine drug screen
   * Positive serum pregnancy test if female
   * Positive ethanol test
7. Clinically significant vital signs

   * Temperature above 100.0 °F
   * Heart rate < 45 or > 100 beats per minute
   * Respiratory rate < 12 or > 20 breaths per minute
   * Systolic blood pressure < 100 or > 140 mm Hg OR diastolic blood pressure < 60 or > 90 mm Hg
8. Known hypersensitivity to any ingredients in the MBX-400 capsules or Placebo capsules (e.g., MBX-400, microcrystalline cellulose, gelatin, titanium dioxide).
9. Scheduled for surgical procedure during the study
10. Investigator deems that subject has a condition that warrants exclusion from or is not suitable for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety | 14 days
  Safety is evaluated by assessing the incidence and severity for 14 days following a single dose of MBX-400 including:
  1. Product-related serious and life-threatening adverse events
  2. Adverse events
  3. Laboratory data abnormalities and clinically significant changes
  4. Electrocardiogram abnormalities and clinically significant changes
  5. Physical exam abnormalities and clinically significant changes
  6. Vital signs abnormalities and clinically significant changes
Area under the plasma concentration-time curve (AUC) | Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, 84 and 96 hours following dosing
  The following pharmacokinetic parameters will be evaluated:
  1. Maximum plasma concentration (Cmax)
  2. Time of maximum plasma concentration (Tmax)
  3. Area under the plasma concentration-time curve (AUC)
  4. Terminal plasma half-life (t1/2)
  5. Apparent plasma clearance (Cl/F)
  6. Apparent volume of distribution (Vd/F)
  7. Amount excreted in urine (Ae)
  8. Urinary clearance (Clu)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Tracey, MD, Principal Investigator — Frontage Clinical Research Center
Locations (1):
- Frontage Clinical Research Center, Hackensack, New Jersey, United States

REFERENCES:
- [Background] Kern ER, Bidanset DJ, Hartline CB, Yan Z, Zemlicka J, Quenelle DC. Oral activity of a methylenecyclopropane analog, cyclopropavir, in animal models for cytomegalovirus infections. Antimicrob Agents Chemother. 2004 Dec;48(12):4745-53. doi: 10.1128/AAC.48.12.4745-4753.2004. PMID 15561852
- [Background] Zhou S, Zemlicka J, Kern ER, Drach JC. Fluoroanalogues of anti-cytomegalovirus agent cyclopropavir: synthesis and antiviral activity of (E)- and (Z)-9-[2,2-bis(hydroxymethyl)-3-fluorocyclopropylidene]methyl-adenines and guanines. Nucleosides Nucleotides Nucleic Acids. 2007;26(3):231-43. doi: 10.1080/15257770701257210. PMID 17454732
- [Background] Mhaske SB, Ksebati B, Prichard MN, Drach JC, Zemlicka J. Phosphonate analogues of cyclopropavir phosphates and their E-isomers. Synthesis and antiviral activity. Bioorg Med Chem. 2009 Jun 1;17(11):3892-9. doi: 10.1016/j.bmc.2009.04.020. Epub 2009 Apr 17. PMID 19410465
- [Background] Li C, Gentry BG, Drach JC, Zemlicka J. Synthesis and enantioselectivity of cyclopropavir phosphates for cellular GMP kinase. Nucleosides Nucleotides Nucleic Acids. 2009 Sep;28(9):795-808. doi: 10.1080/15257770903172720. PMID 20183619
- [Background] Gentry BG, Gentry SN, Jackson TL, Zemlicka J, Drach JC. Phosphorylation of antiviral and endogenous nucleotides to di- and triphosphates by guanosine monophosphate kinase. Biochem Pharmacol. 2011 Jan 1;81(1):43-9. doi: 10.1016/j.bcp.2010.09.005. Epub 2010 Sep 22. PMID 20846508
- [Background] Chou S, Bowlin TL. Cytomegalovirus UL97 mutations affecting cyclopropavir and ganciclovir susceptibility. Antimicrob Agents Chemother. 2011 Jan;55(1):382-4. doi: 10.1128/AAC.01259-10. Epub 2010 Nov 1. PMID 21041510
- [Background] James SH, Hartline CB, Harden EA, Driebe EM, Schupp JM, Engelthaler DM, Keim PS, Bowlin TL, Kern ER, Prichard MN. Cyclopropavir inhibits the normal function of the human cytomegalovirus UL97 kinase. Antimicrob Agents Chemother. 2011 Oct;55(10):4682-91. doi: 10.1128/AAC.00571-11. Epub 2011 Jul 25. PMID 21788463